CLINICAL TRIAL: NCT05593029
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of the Safety and Efficacy of Flexible Doses of SEP-363856 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder
Brief Title: A Trial of the Safety and Efficacy of SEP-363856 in the Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 382-201-00001
Record Dates: First submitted 2022-10-10; First posted 2022-10-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: MDD; SEP-363856; Antidepressant Therapy; ADT; Depression; Depressive Disorder; Major Mood Disorders; Mental Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Mental Disorders | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEP-363856 & ADT (Antidepressant Therapy) (Experimental)
  Interventions: Drug: SEP-363856
- Placebo & ADT (Antidepressant Therapy) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SEP-363856 — Tablet
  Arms: SEP-363856 & ADT (Antidepressant Therapy)
Other: Placebo — Placebo
  Arms: Placebo & ADT (Antidepressant Therapy)

SUMMARY:
Demonstrate ability of SEP-363856 to be superior to placebo as an adjunctive therapy to ADT in change from baseline in depressive symptoms (MADRS & CGI-S) in MDD patients who had an inadequate response to prior ADT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects between 18-65 years of age, with a primary diagnosis of major depressive disorder and in a current major depressive episode
* Current major depressive episode must be at least 8 weeks and no longer than 2 years in duration
* History of an inadequate response to at least 1 and no more than 3 antidepressant treatments in the current major depressive episode

Exclusion Criteria:

* Subjects who report an inadequate response to more than 3 antidepressant treatments in the current episode
* Subjects with a lifetime history of schizophrenia spectrum or other psychotic disorder, bipolar or related disorder, major or mild neurocognitive disorder, neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent/ follow study directions/ or otherwise safely participate in the study, borderline or antisocial personality disorder.
* Subjects with a current diagnosis of post-traumatic stress disorder, obsessive compulsive disorder, panic disorder, or eating disorder (including anorexia nervosa or bulimia).
* Sexually active subjects, who could become pregnant, not agreeing to practice 2 sponsor approved methods of birth control or remain abstinent during the trial and for 30 days (females) or 90 days (males) after last dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS) | From baseline to week 14
  Change from the baseline to the Montgomery Åsberg Depression Rating Scale (MADRS) total score.
  The Montgomery Åsberg Depression Rating Scale consists of 10 items, each rated from 0 to 6 (for a total score of 0 to 60). A higher score represents a higher severity of the level of depression.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity of Illness (CGI-S) | From baseline to week 14
  Change from baseline in the Clinical Global Impression - Severity of Illness (CGI-S).
  Clinical Global Impression - Severity of Illness will be measured on a scale from 1-7 where a higher score represents a higher severity of disease.

CONTACTS AND LOCATIONS:
Locations (77):
- United States (53):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scottsdale Clinical Research, Scottsdale, Arizona
  - DelSol Research, Tucson, Arizona
  - Pillar Clinical Research, Bentonville, Arkansas
  - ProScience Research Group, Culver City, California
  - Wr-Pri, Llc, Encino, California
  - Collaborative NeuroScience Research , LLC, Garden Grove, California
  - Alliance Research, Long Beach, California
  - ATP Clinical Research, Inc., Orange, California
  - Anderson Clinical Research, Redlands, California
  - California Mental Behavioral Health, Santee, California
  - Schuster Medical Research Institute SMRI, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Collaborative Neuroscience Research LLC, Torrance, California
  - Sunwise Clinical Research with is in Lafayette, CA, Walnut Creek, California
  - Institute of Living Hartford Hospital, Hartford, Connecticut
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - K2 Medical Research, Maitland, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Clinical Neuroscience Solutions Inc. dba CNS Healthcare, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - K2 Medical Research, Tampa, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - Renew Health Clinical Research, Snellville, Georgia
  - MetroMed Clinical Trials, Chicago, Illinois
  - AMR Convention Research, Warrenville, Illinois
  - Benchmark Research, Shreveport, Louisiana
  - Cenexel CBH (CBH Health), Gaithersburg, Maryland
  - Copley Clinical, Boston, Massachusetts
  - Boston Clinical Trials, Roslindale, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Vitalix Clinical, Worcester, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Integrative Clinical Trials, Brooklyn, New York
  - Basil Clinical, Inwood, New York
  - Berman Clinical, New York, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Patient Priority Clinical Studies LLC, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Suburban Research Associates, West Chester, Pennsylvania
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Donald J. Garcia, Jr., MD, PA, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - DM Clinical Research - Belliare, Houston, Texas
  - Psychiatric And Behavioral Solutions, LLC, Millcreek, Utah
  - Core Clinical Research, Everett, Washington
- Bulgaria (5):
  - Diagnostic Consultive Center Higya AD, Pazardzhik
  - Ambulatory for Group Practice for Specialized Psychiatrics Help PHILIPOPOLIS OOD, Plovdiv
  - Medical Center Sveti Naum, Sofia
  - DCC-Mladost M OOD, Varna
  - Mental Health Center Vratsa, Vratsa
- Canada (3):
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Institute of Mental Health Research IMHR, Ottawa, Ontario
  - Centre for Addiction and Mental Health (CAMH & University of Toronto), Toronto, Ontario
- Czechia (4):
  - BRAIN-SOULTHERAPY s.r.o., Kladno, Central Bohemia
  - A-Shine s.r.o., Ptzen, Plzeň Region
  - National Institute of Mental Health, Klecany
  - Clintrial s.r.o., Prague
- Germany (5):
  - Velocity Clinical Research Wiesbaden, Wiesbaden, Hesse
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Chemnitz, MA
  - Private Practice Kusserow, Stralsund, Mecklenburg-Vorpommern
  - Somni Bene Institut for Medical Research, Schwerin, Mecklenburg
  - Arztepartnerschaft Dr. med. J. Springhub/ W. Schwarz-Studienzentrum Nord-West, Westerstede
- Hungary (2):
  - ClinExpert Kft., Budapest
  - Semmelweis University, Budapest
- Poland (5):
  - Praktyka Lekarska Malgorzata Wojtanowska-Bogacka, Poznan, Greater Poland Voivodeship
  - Osrodek Badan Klinicznych CLINSANTE, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MlynowaMed - Bialystok, Bialystok, OH
  - Centrum Medyczne Luxmed Sp.z. o.o., Lublin
  - Indywidualna SpecjalistycznaPraktyka Lekarska AgnieszkaRemlinger-Molenda, Szkolkarska 32

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com